CLINICAL TRIAL: NCT05648682
Title: Comparison of the Effectiveness of Three Different Gargates in Radiotherapy-Associated Oral Mucositis Management in Head and Neck Cancer Patients: A Randomized Controlled Study
Brief Title: Comparison of the Effectiveness of Three Different Gargates in Radiotherapy-Associated Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Zeynep Yilmaz, Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBU_RKC
Record Dates: First submitted 2022-11-25; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancers; Oral Mucositis
Keywords: nurse; radiotherapy; salin; sodium bicarbonate; thyme honey; Head and Neck Cancers; Oral Mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline (Experimental): The patients in the group gargling with saline were given in a 500 ml bottle at each visit for one week of use. Patients were told that they should gargle using approximately two tablespoons of the solution given for each usage.
  Interventions: Other: Salin
- Sodium Bicarbonate (Experimental): The sodium bicarbonate solution prepared by the researcher by mixing one teaspoon of baking soda (4.5 grams) into 500 ml of distilled water by the researcher was given to the patients in the group gargling with sodium bicarbonate for a one-week use at each interview. Patients were told that they should gargle using approximately two tablespoons of the solution given for each usage.
  Interventions: Other: Sodium bicarbonate
- Thyme Honey (Experimental): 20 ml of honey was diluted in 100 ml distilled water bottles by the researcher to the patients in the group gargling with thyme honey. For a week's use, the patient was given five honey solutions in 100 ml bottles at one time at each visit. Patients were told that they should gargle using approximately two tablespoons of the solution given for each use.
  Interventions: Other: Thyme honey
- Control (Experimental): No solution was given to the patients in the control group by the researcher.
  Interventions: Other: Control

INTERVENTIONS:
Other: Salin — Patients were told that they should gargle using approximately 2 tablespoons of the solution given for each use. SF solution was obtained from the medical company as 500 ml separately for each patient.
  Arms: Saline
Other: Sodium bicarbonate — Patients were told that they should gargle using approximately two tablespoons of the solution given for each use. The 500 ml distilled water bottle to be used for the SB solution was obtained from the medical company, separately for each patient.
  Arms: Sodium Bicarbonate
Other: Thyme honey — Patients were told that they should gargle using approximately 2 tablespoons of the solution given for each use.
  Arms: Thyme Honey
Other: Control — The patients continued to use the antifungal solution containing the active ingredient nystatin, which was prescribed routinely in the clinical procedure, 3 times a day.
  Arms: Control

SUMMARY:
This study was conducted to compare the effectiveness of thyme honey, saline and sodium bicarbonate solution in the management of oral mucositis in patients with head and neck cancer receiving radiotherapy.

DETAILED DESCRIPTION:
The research was conducted as a randomized controlled clinical trial between January 2020 and January 2022. The sample of the research; Patients who applied to Hospital Radiotherapy Unit, received 50-60 Gy radiotherapy in the oral cavity, had a primary diagnosis of head and neck cancer, had no metastasis, had no complaints about mucositis, were older than 18 years old, spoke Turkish, and agreed to participate, in the study. With the closed-envelope randomization method, 48 patients were included in the sample, 12 patients for each of the saline, sodium bicarbonate, thyme honey, and control groups. The routine protocol of the clinic was applied to the control group. Patients in the intervention group (thyme honey, saline and sodium bicarbonate group) were treated 3 times a day for 6 weeks, in addition to the routine protocol of the clinic; they were asked to gargle with 20 ml of the solution in the group they were randomized to, 15 minutes before, 15 minutes and 6 hours after radiotherapy. Intraoral evaluations were made every week by the responsible physician of the radiotherapy unit, who did not know which group the patients were in (single blind). Study data; Obtained using the Sociodemographic and Disease Data Collection Form, the National Cancer Institute Common Toxicity Criteria v4.03, the Oral Evaluation Guide, and the Washington University Quality of Life Questionnaire. In the study, Chi-square analysis was used for the relationship between two categorical variables, One-way Anova for differences in measurements, Levene test for homogeneity of variance, and Bonferroni analysis to find out from which group or groups the difference originated. Support was received from the Health Sciences University Scientific Research Project Office for the study (2020/029)

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis is head and neck cancer
* To be receiving radiotherapy at a dose of 50-60 Gy in the oral cavity
* Not be metastatic
* OM grade 1 (according to NCI-CTCAE v4.03)
* Be 18 years or older
* Volunteer to participate in the study
* Speak Turkish

Exclusion Criteria:

* Have an autoimmune disease
* Have dental disease
* Using dentures
* Being allergic to thyme honey
* Refusing to participate in the research
* To have received radiotherapy treatment in the 6-month period before the start of the study

Criteria for terminating the study

* The patient's desire to leave the study
* Continuing the treatment in another city
* Interruption or termination of radiotherapy treatment
* Patient's death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=6 patients have oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change= 12 patients have oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of control group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of saline group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of sodium bicarbonate group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=8 patients have oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of thyme honey group patients with oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=6 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have Grade 1-2 oral mucositis 8 patients have Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=7 patients have Grade 1-2 oral mucositis 5 patients have Grade 3 oral mucositis
Number of control group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have Grade 1-2 oral mucositis 8 patients have Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=10 patients have Grade 1-2 oral mucositis 2 patients have Grade 3 oral mucositis
Number of saline group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have Grade 1-2 oral mucositis
  1 patient has Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=4 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have Grade 1-2 oral mucositis
  1 patient has Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=7 patients have Grade 1-2 oral mucositis 5 patients have Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=7 patients have Grade 1-2 oral mucositis 5 patients have Grade 3 oral mucositis
Number of sodium bicarbonate group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=10 patients have Grade 1-2 oral mucositis 2 patients have Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Week 0
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | First week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=0 patient has Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Second week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=8 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Third week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fourth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have Grade 1-2 oral mucositis
  1 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Fifth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=11 patients have Grade 1-2 oral mucositis
  1 patient has Grade 3 oral mucositis
Number of thyme honey group patients with severe oral mucositis assessed by National Cancer Institute Criteria For Adverse Events v4.03 (NCI-CTCAE v4.03) | Sixth week of radiotherapy
  National Cancer Institute Criteria For Adverse Events v4.03 is used to determine the severity of OM due to radiotherapy. The severity of OM is graded from 0 to 5. Grade 0 means no mucositis. Grade 1 has mucositis but no complaints or mild mucositis. There are mild ulcerations in the mouth. Grade 2 has enlarged ulcerated areas with moderately painful mucositis that does not interfere with food intake but requires a change of type. Grade 3 has severely painful mucositis and large ulcerated areas with bleeding that interfere with food intake. Grade 4 is classified as mucositis requiring immediate medical intervention and Grade 5 is death due to mucositis.
  Change=12 patients have Grade 1-2 oral mucositis 0 patient has Grade 3 oral mucositis
Control group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Week 0
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=83,57
Control group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Second week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=73,71
Control group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Fifth week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=65,30
Saline group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Week 0
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=82,99
Saline group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Second week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=69,67
Saline group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Fifth week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=65,30
Sodium bicarbonate group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Week 0
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=75,31
Sodium bicarbonate group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Second week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=62,17
Sodium bicarbonate group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Fifth week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=52,56
Thyme honey group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Week 0
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=85,59
Thyme honey group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Second week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=73,71
Thyme honey group patients' quality-of-life scores as assessed by The University of Washington Quality of Life Questionnaire | Fifth week of radiotherapy
  The 12 items included in the University of Washington Quality of Life Questionnaire question are "pain, appearance, activity, fun, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety". In its scoring, each of the answers to the 12 items is scored from 0 (worst quality of life) to 100 (the best quality of life). In each item, the worst answer is scored as "0", while the best answer is scored as "100".
  Change=70,42

CONTACTS AND LOCATIONS:
Overall Officials: Fatma İlknur ÇINAR, Study Director — Saglik Bilimleri Universitesi; Zeynep YILMAZ, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Zeynep YILMAZ, Bilecik, Turkey (Türkiye)